CLINICAL TRIAL: NCT05477966
Title: A Retrospective Cohort Study to Develop Markers for TB Severity and Treatment Progress
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jae-Joon Yim (Other)
Responsible Party: Sponsor-Investigator, Jae-Joon Yim, Principal Investigator, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: H-2206-179-1336
Record Dates: First submitted 2022-07-18; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Tuberculoses; Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medical records review — The clinical characteristics at the time of diagnosis of rifampin-susceptible pulmonary tuberculosis patients, the Xpert MTB/RIF assay Ct value, the tuberculosis activity score based on AI of the chest image, and treatment results will be collected retrospectively through medical records.

SUMMARY:
The objective of this study is to compare how accurately the Xpert MTB/RIF assay Ct value at diagnosis and the AI-based tuberculosis activity score predict the treatment outcome of rifampin-susceptible pulmonary tuberculosis patients. As a retrospective observational study, data from patients diagnosed with rifampin susceptible pulmonary tuberculosis through the Xpert MTB/RIF assay performed on sputum in 2019 at the participating institutions will be analyzed (up to 900 people).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rifampin-susceptible pulmonary tuberculosis by Xpert MTB/RIF assay with sputum samples between January 1, 2019 and December 31, 2019

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 900 patients diagnosed with rifampin-susceptible pulmonary tuberculosis through the Xpert MTB/RIF assay performed on sputum between January 1, 2019 and December 31, 2019 at the participating institutions
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-07-18 (Estimated); Primary Completion 2023-07-18 (Estimated); Study Completion 2023-07-18 (Estimated)

PRIMARY OUTCOMES:
Negative culture conversion until 8 weeks after initiation of treatment | Within 8 weeks of initiating treatment
  Conversion from positive tuberculosis culture to negative tuberculosis culture
Time to negative culture conversion | Within 6 months of initiating treatment
  Time (days) to conversion from positive tuberculosis culture to negative tuberculosis culture
Treatment outcome including 1) Cure 2) Treatment completion 3) Treatment failure 4) Death 5) Loss of follow-up 6) Unknown | Within 2 years of initiating treatment
  1. Cure: confirmed negative culture conversion plus negative culture results from at least one sputum on the month of treatment completion
  2. Treatment completion: confirmed negative culture conversion at least once during treatment
  3. Treatment failure: positive culture results after 4 months of treatment
  4. Death: death during treatment
  5. Loss of follow-up: loss of follow-up during treatment
  6. Unknown

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.